CLINICAL TRIAL: NCT06449430
Title: Randomized Clinical Trial of the Use of Propofol as a Sedative Agent Versus Spinal Analgesia With Bupivacaine in External Cephalic Version
Brief Title: Use of Propofol as a Sedative Agent Versus Spinal Analgesia With Bupivacaine in External Cephalic Version
Acronym: PropoSpinECV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMIB-ECV-2024-01
Record Dates: First submitted 2024-05-28; First posted 2024-06-10 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications | interventions — Propofol; Bupivacaine

STUDY DESIGN:
Intervention Model Description: An open randomized clinical trial has been designed comparing sedation with propofol versus spinal analgesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedation with propofol (Experimental): Atropine 0.4 mg intravenous bolus and intravenous propofol will be administered through a continuous infusion with a target plasma concentration between 4-6 micrograms/mL maintaining a BIS between 65-75, following the protocol used by Sánchez-Romero J et al. (doi:10.3390/jcm11030489). For this, an intravenous infusion pump (Agilia SP TIVA ES, Fresenius Kabi AG, Bad Homburg, Germany) will be used. After the administration of propofol, a period of 3 minutes will be waited before starting the procedure to ensure the target plasma concentration.
  Interventions: Drug: Sedation with propofol
- bupivacaine (Active Comparator): A combined spinal-epidural anesthesia technique will be performed with a spinal dose of 5-7.5 mg of hyperbaric bupivacaine and 20 μg of intrathecal fentanyl, along with the placement of an epidural catheter, following the protocol used by Brogly N et al. in "Protocols of the Obstetric Anesthesia Section of SEDAR, 2021". After the administration of epidural anesthesia, a period of 3 minutes will be waited before starting the procedure to ensure effective anesthesia.
  Interventions: Drug: Spinal analgesia with bupivacaine

INTERVENTIONS:
Drug: Sedation with propofol — Sedation with propofol
  Arms: Sedation with propofol
Drug: Spinal analgesia with bupivacaine — Spinal analgesia with bupivacaine
  Arms: bupivacaine

SUMMARY:
External Cephalic Version (ECV) is a maneuver to modify fetal position in pregnant women with a non-cephalic presentation. Its objective is to achieve a cephalic presentation that allows for vaginal delivery with less risk than a vaginal breech delivery or a cesarean section. ECV is an effective technique to reduce the rate of cesarean sections and is recommended by the Spanish Society of Obstetrics and Gynecology (SEGO) and the World Health Organization (WHO) Cesarean Section Working Group. The WHO aims to reduce interventionism in childbirth globally and implement non-clinical measures to reduce the rate of unnecessary cesarean sections.

Despite Propofol is a sedative agent commonly used by anesthesiologist in countless ambulatory procedures in obstetric anaesthesia, it has been little studied in ECV, and its effect has not been compared with other commonly used agents such as remifentanil or spinal analgesia. The Obstetric Anesthesiology Section of the Spanish Society of Anesthesiology and Resuscitation recommends the use of locoregional analgesia in ECV.

DETAILED DESCRIPTION:
This project involves a randomized clinical trial to compare the effect of sedation with propofol versus spinal analgesia in ECV. Therefore, the objectives of this study are:

* To compare the effect of sedation with Propofol on the success rate of ECV compared to spinal analgesia.
* To compare the effect of sedation with Propofol on the rate of complications of ECV compared to spinal analgesia.
* To compare the effect of sedation with Propofol on the length of hospital stay of ECV compared to spinal analgesia.

Locoregional analgesia requires a longer hospital stay than sedation with Propofol and may mask an early diagnosis of complications after ECV, such as placental abruption, which is identified in the initial stages by intense abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation.
* Older than 18 years.
* Non-cephalic presentation.
* Desire to attempt a vaginal birth.
* Normal blood count and coagulation prior to the intervention

Exclusion Criteria:

* Age under 18 years old.
* Multiple gestation.
* Cephalic presentation.
* Risk of fetal compromise.
* Unexplained active bleeding.
* Absolute contraindication for vaginal delivery (Placenta Previa)
* 2 or more previous cesarean sections.
* Previous myomectomy with entry into the uterine cavity
* Maternal fever.
* Thrombocytopenia (<85,000 platelets).
* Maternal spinal anomaly.
* Intolerance or allergy to Propofol or any of its components.
* Intolerance or allergy to bupivacaine or any of its components.
* Contraindication for intrathecal sedation or analgesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 270 (Estimated)
Dates: Start 2024-07-06 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
compare the success rate of external cephalic version | Up to 24 months.
  Number of external cephalic version when Propofol is used as a sedative agent or spinal analgesia.

SECONDARY OUTCOMES:
ECV (external cephalic version) complication rate when using Propofol as a sedative agent or spinal analgesia. | Up to 24 months.
  Number of complications
rate of emergency cesarean sections in the first 24 hours after the procedure when using Propofol as a sedative agent or spinal analgesia in ECV. | Up to 24 months
  Number of emergency cesarean
postprocedural pain when Propofol is used as a sedative agent or spinal analgesia in ECV | Up to 24 months
  Visual Analogue Scale (VAS) pain consists of 9 items on which participants rate their perceived dizziness on a scale between 1 (no dizziness) and 10 (most dizziness) in different visual vertigo-inducing environments
rate of clinically relevant hypotension (SBP <90 mmHg or a 20% decrease from baseline SBP) when using Propofol as a sedative agent or spinal analgesia in ECV | Up to 24 months
  number of episodes of hypotension hypotension
rate of nausea or vomiting when using Propofol as a sedative agent or spinal analgesia in ECV. | Up to 24 months
  Level of nausea or vomiting in clinical history
angle of progression of fetal presentation as a predictor of ECV success. | Up to 24 months
  angle of progression of fetal presentation
angle of progression of fetal presentation as a predictor of complications of ECV. | Up to 24 months
  angle of progression of fetal presentation as a predictor of complications of ECV.
degree of tissue oxygenation of the placenta during ECV by analyzing a pilot sample with infrared spectroscopy (NIRS) | Up to 24 months
  degree of tissue oxygenation

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sanchez-Romero J, Falcon-Arana L, Blanco-Carnero JE, Garcia-Ferreira J, Herrera-Gimenez J, Fuentes-Garcia D, Araico-Rodriguez F, Gallego-Pozuelo RM, Nieto-Diaz A, de Paco-Matallana C. Randomized clinical trial of the use of Propofol as a sedative agent versus spinal analgesia with bupivacaine in External Cephalic Version (PropoSpinECV): study protocol for a randomized clinical trial. Trials. 2025 Oct 9;26(1):398. doi: 10.1186/s13063-025-09105-0. PMID 41068932